CLINICAL TRIAL: NCT06202170
Title: The Validity and Reliability of the 30-Second Fast-Paced Walk Test in Patients With Total Knee Arthroplasty
Brief Title: Validity and Reliability of 30SFPW Test Patients With TKA
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Ozcan, Msc. Pt, Dokuz Eylul University
Other Study IDs: 6748-GOA
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty, knee, 30-Second Fast-Paced Walk Test, validity, reliability.
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Walking speed after total knee arthroplasty (TKA) can be used as a simple tool to monitor postoperative recovery. There are different protocols for gait assessment in patients with TKA. The 30 Second Fast Walk Test (30SFW) is a simple, low-cost and easy-to-apply assessment method that requires very little equipment in clinical settings. 30SFW is a reliable, valid test of walking ability in patients with knee osteoarthritis (OA).

Objective: To investigate the reliability and validity of the 30SFW test in the evaluation of gait in patients with TKA.

ELIGIBILITY:
Inclusion Criteria:patients who had primary TKA surgery at least six months ago, being diagnosed with preoperative knee OA, and volunteering to participate in the research -

Exclusion Criteria:had a previous orthopedic, neurological, or systemic disease that effects walking or standing, body mass index of 40 kg / m2 and over, having any other surgery on the same limb that effect walking, and revision TKA.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who had primary TKA surgery at least six months ago
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
30SFPWT | 1 Hour-30 Seconds
  30 Second Fast-Paced Walk Test

SECONDARY OUTCOMES:
Hss Knee Socre | 15 minutes
SF-12 Quality Life Score | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No